CLINICAL TRIAL: NCT03058887
Title: Investigating the Effectiveness and Feasibility of Exercise on Microcirculatory Parameters and Quality of Life in Systemic Sclerosis Patients Experiencing Raynaud's Phenomenon.
Brief Title: The Effects of Exercise in Patients With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAS: 68096
Record Dates: First submitted 2016-10-13; First posted 2017-02-23 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Systemic Sclerosis; Raynaud's Phenomenon; Quality of Life
Keywords: High Intensity Interval Training; Exercise; Microcirculation
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm cranking (Experimental): exercising for 3 months twice per week.
  Interventions: Other: Exercise intervention - arm cranking
- Cycling (Experimental): exercising for 3 months twice per week.
  Interventions: Other: Exercise intervention - Cycling
- Control group (No Intervention): No exercise intervention.

INTERVENTIONS:
Other: Exercise intervention - Cycling — The patients that will be randomly allocated to the exercise group - cycling will be requested to perform an exercise session on a cycle ergometer. Each training will be consisted of high intensity interval training for 30 minutes (30s 100% PPO/ 30s passive recovery) twice per week for 3 months. Patients will perform two visits for the baseline measurements prior the exercise intervention by repeating them at the end of the exercise intervention (follow up measurements).
  Arms: Cycling
Other: Exercise intervention - arm cranking — The patients that will be randomly allocated to the exercise group - arm cranking will be requested to perform an exercise session on an arm crank ergometer. Each training will be consisted of high intensity interval training for 30 minutes (30s 100% PPO/ 30s passive recovery) twice per week for 3 months. Patients will perform two visits for the baseline measurements prior the exercise intervention by repeating them at the end of the exercise intervention (follow up measurements).
  Arms: Arm cranking

SUMMARY:
Systemic sclerosis (SSc) is a multisystem connective tissue disease characterised by vascular abnormalities and fibrosis, including those of the skin and can be categorised as either Limited cutaneous scleroderma or Diffuse cutaneous scleroderma. It is estimated that more than 90% of patients with SSc experience Raynaud's phenomenon (RP) at regular intervals during the course of their disease. Approximately 50% of patients with SSc develop severe digital ischaemia and/or ulceration which seems to be painful, difficult to heal, susceptible to infections and heavily influences quality of life and increases SSc-related disability.

Medical treatment is commonly used as an effective first line approach in the NHS policy when uncontrolled RP attacks emerge. However, considering the short-term side effects (oedema, headaches, heart palpitations, dizziness and constipation) but also the long-term side effects of nifedipine (heart dysfunction and increased cardiovascular risk) as well as the financial cost of this approach, alternative approaches with less side effects and less cost implications are warranted.

An alternative approach would be to implement a programme of therapeutic exercise that would be suitable for this patient group. To the investigators knowledge the efficacy of exercise on microcirculation in RP has not been previously examined. In this regard, high intensity interval training (HIIT) has come to prominence over the last years for its effectiveness in inducing greater improvements in vascular function than moderate intensity continuous training. Due to the variation in HIIT protocols evidence is limited to support which protocol is the most effective in SSc patients. Moreover, it should be noted that the chief aim of the research project is to encourage long-term adherence to physical activity and rehabilitation programmes in these patients which might be beneficial for the vascular function. A short HIIT protocol (30seconds/passive recovery) may elicit more favourable patient reported satisfaction /enjoyment levels compared to other longer exercise duration protocols. A short HIIT protocol (30seconds/passive recovery) has demonstrated to be well tolerated, preferred protocol with a low perception of effort, patient comfort and with a longer time spent at high percentage of V̇O2peak than a longer HIIT protocol with active recovery phases in chronic heart failure patients. More recent evidence supports this notion; when enjoyment levels in an overweight/obese cohort were examined after a short HIIT protocol.

Although it is known that HIIT is capable to improve vascular function and potentially the microcirculatory parameters, evidence is scarce regarding the mode of exercise that will be more effective on digital microcirculation where the RP attacks are present in SSc patients. Assumptions could be made that utilising an upper-body exercise would potentially be more beneficial for the digital microcirculation rather than lower-body exercise where the working muscles promote the blood flow in the lower limbs. Hence, the differential effects that may occur by the upper- and lower-limb exercise on the digital microcirculation in SSc patients should be examined.

Resistance training (RT) alone has shown significant improvements in the function of the vasculature; moreover, a combination of aerobic and RT have shown both in the past and recently important enhances in the vascular function and microcirculation. However, the limited number of studies have investigated the effects of RT on vasculature bespeaks a lack of concrete evidence. Moreover, to the investigators knowledge the effects of combined exercise (RT and aerobic exercise) utilising a HIIT protocol and RT on microcirculation has yet to be examined.

Aims:

The primary aim of the present study is to examine the feasibility of exercise in patients with Systemic Sclerosis experiencing Raynaud's Phenomenon.

ELIGIBILITY:
Inclusion criteria

* Patients diagnosed with Limited Cutaneous Systemic Sclerosis according to the 2013 ACR/EULAR criteria experiencing Raynaud's phenomenon.
* Men or women aged 18-80 years old.
* Disease duration between 1 to 10 years.
* Patients should be able to perform exercise. Exclusion criteria
* Patients with advanced pulmonary arterial hypertension or interstitial lung disease.
* Patients who are diagnosed with another inflammatory condition.
* Patients presenting myositis with proximal muscle weakness.
* Patients with New York Heart Association class 3 or 4.
* Current smokers or people who stopped smoking within 4 weeks of health screening.
* Women who are currently pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Part I (Pilot study): Microcirculation in the digital area | 12 months
  Microcirculation will be assessed via the combination of iontophoresis and laser doppler fluximetry in order to assess the microvascular reactivity pre and post the exercise intervention in the digital area.
Part II (Feasibility study): Feasibility of a combined exercise protocol (aerobic with resistance training). | 12 months
  The feasibility of the exercise protocol will be assessed via the acceptability of the exercise protocol which will be measured with certain questionnaires (task self efficacy, enjoyment levels and engagement levels), individual experiences from the exercise sessions (interviews) and compliance criteria (e.g. completion of > 75% of the scheduled sessions and/or percentage of dropouts).
  All these measures will be aggregated in order to conclude whether a combined exercise is feasible to be implemented in patients with systemic sclerosis.
Part II (Feasibility study): Assessment of Quality of life | 12 months
  The quality of life will be assessed through a modified version of EQ-5D-5L questionnaire, a 6 minute-walking test that will assess the functional capacity to perform daily activities and individual experiences (interviews).

SECONDARY OUTCOMES:
Part I (Pilot study): Quality of life | 12 months
  The quality of life will be assessed through a modified version of EQ-5D-5L questionnaire, a 6 minute-walking test that will assess the functional capacity to perform daily activities and individual experiences (interviews).
Part I (Pilot study): Enjoyment levels and acceptability of exercise | 12 months
  The acceptability of the exercise protocol and enjoyment levels which will be assessed via certain questionnaires (task self efficacy, enjoyment levels and engagement levels)
Part II (Feasibility): Microcirculation in the digital area | 12 months
  Microcirculation will be assessed via the combination of iontophoresis and laser doppler fluximetry in order to assess the microvascular reactivity pre and post the exercise intervention in the digital area.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Sheffield Hallam University, Sheffield
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Mitropoulos A, Gumber A, Crank H, Akil M, Klonizakis M. Exploring the feasibility of an exercise programme including aerobic and resistance training in people with limited cutaneous systemic sclerosis. Clin Rheumatol. 2020 Jun;39(6):1889-1898. doi: 10.1007/s10067-019-04921-7. Epub 2020 Jan 14. PMID 31933034
- [Derived] Mitropoulos A, Gumber A, Akil M, Klonizakis M. Exploring the microcirculatory effects of an exercise programme including aerobic and resistance training in people with limited cutaneous systemic sclerosis. Microvasc Res. 2019 Sep;125:103887. doi: 10.1016/j.mvr.2019.103887. Epub 2019 Jun 17. PMID 31220505
- [Derived] Mitropoulos A, Gumber A, Crank H, Akil M, Klonizakis M. Investigating the effectiveness and feasibility of exercise on microvascular reactivity and quality of life in systemic sclerosis patients: study protocol for a feasibility study. Trials. 2018 Nov 21;19(1):647. doi: 10.1186/s13063-018-2980-1. PMID 30463598
- [Derived] Mitropoulos A, Gumber A, Crank H, Akil M, Klonizakis M. The effects of upper and lower limb exercise on the microvascular reactivity in limited cutaneous systemic sclerosis patients. Arthritis Res Ther. 2018 Jun 5;20(1):112. doi: 10.1186/s13075-018-1605-0. PMID 29871697